CLINICAL TRIAL: NCT05381987
Title: The Effectiveness of Radial Shockwave Therapy on Myofascial Pain Syndrome: A Mixed Method Study That Combines a Randomised Control Trial and Semi-Structured Interview.
Brief Title: The Effectiveness of Radial Shockwave Therapy on Myofascial Pain Syndrome in Neck and Upper Back.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RAC# 2221047
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2022-05

CONDITIONS: Myofascial Pain Syndrome of Neck
Keywords: Myofascial pain syndrome, trigger point pain, shockwave, randomised controlled trial
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Intervention Model Description: This study will make use a pragmatic, two-arm, parallel, doubled-blind, randomised controlled as the study design.
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomisation allocation sequence will be based on computer-generated random sequence using permuted block size of 4 and concealed random allocation using sealed opaque envelopes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (experimental) group (Experimental): These will receive a total of 6 sessions with a week's interval of radial shockwaves that will be performed using a (Storz Medical) device with the following manufacturer's parameters: 0.57mJ/mm2 (intensity 1.5 bar) applied as low energy, pulses 2000, frequency 15 Hz. The D20 transmitter (Ø 20 mm) headpiece will be used. Total treatment time including standard PT stretches and exercises would be 30 minutes). The radial shockwave will be delivered by designated physiotherapist, who will evaluate the participants before the treatment. Before the treatment, the treating physical therapist would ensure aseptic techniques, they would ensure the participants skin is intact and clean coupling gel will be used during the treatment. Furthermore prior to treatment, the myofascial triggers would be specifically confirmed by twitching response induced by a localized probe using a digital algometer.
  Interventions: Device: Radial shockwave therapy
- Control (placebo) group (Placebo Comparator): These will receive an identical treatment regime except that they will receive a none-therapeutic level energy shock of 0.03 mJ/mm2, an ineffective (a non-therapeutic) level of radial shockwave therapy, and participants will be blinded to their treatment by only hearing the sound from the shockwave machine.
  Interventions: Device: Radial shockwave therapy

INTERVENTIONS:
Device: Radial shockwave therapy — Shockwave Storz Medical device, Doulith SD1, Tower (BT)
  Other Names: Shockwave Storz Medical device, Doulith SD1, Tower (BT)

SUMMARY:
Introduction: Myofascial pain syndrome (MPS) is a common, costly and often persistent musculoskeletal problem. Radial shockwave (RSW) is one of the most common treatment for MFS. However, a recent systematic review found very low-level evidence to support its short-term benefit, due to poor methodological qualities. The authors therefore recommended further large scale, good quality placebo-controlled trials (RCT) in this area. Further still, previous studies have not considered the experiences of patient regarding this intervention.

Study Objectives: To determine the effectiveness of RSW compared to placebo for the treatment of patients with MPS in neck and upper back, and to establish the experiences of patients receiving the treatment.

Research Questions: Is RSW therapy more effective at improving MPS compared to a placebo? What are the experiences of patients with MPS receiving this treatment?

Methods: A pragmatic double blind RCT to investigate the effectiveness of RSW on patients with MPS and a semi-structured-interview to investigate the patients' experience of receiving the treatment.

Sample: 120 potential participants with MPS for the RCT and 20 participants for the semi-structured qualitative interview.

Interventions: The Intervention group will receive a total of 6 sessions of RSW following manufacturer's parameters: 1.5 bar, pulses 2000, frequency 15 Hz (Time 3 minutes). The Control group will receive an identical treatment except that the they will receive a no energy shock of 0.3 bar, frequency 15 and no pulses.

Outcome measures: Improvements in the patient's numeric pain scale (NPS), neck disability index (NDI), pressure pain threshold (PPT) and SF-12 questionnaires at 4, 8 and 12 weeks' follow-up between the two groups.

Significance of the Study's Outcome: The expectation is that this study will add to the body of knowledge required to help patients, healthcare practitioners, policy makers and researchers make effective treatment choices on RSW in the management MFS.

DETAILED DESCRIPTION:
INTRODUCTION Myofascial pain syndrome (MPS) is a common, costly and often persistent musculoskeletal problem that affects 85% of the general population at some point in their lifetime (Fleckenstein et al, 2010; Simon, 1996). Reported overall rates vary between male and female population and with different patient populations. MPS has been reported as the leading cause of chronic and persistent musculoskeletal regional pain such as neck pain, shoulder pain, chronic back pain and facial pain (Li et al, 2017). In the United States, the estimated economic cost for the management of chronic pain is $560-$635 billion per annum for medical care and disability programs, with the potential to increase year on year (Gaskin & Richard, 2012). Therefore, it is important that chronic musculoskeletal pain such as MPS in the neck and upper back is treated efficiently and effectively to improve patient's clinical outcomes and experience.

The clinical manifestation of MPS varies widely because it is not a distinct pathology. It is characterised by localized pain, muscle tenderness, palpable intramuscular taut band, local twitch response, referred pain, muscle spasm and sleep disturbance (Fernández-de-las-Peñas et al, 2012; Sciotti et al, 2001; Alvarez & Rockwell, 2001; Travell & Simmons, 1999). Myofascial trigger points can produce symptoms of pain upon palpation and pressure. A nail bed palpation by pressing manually with a thumb or using a digital algometer probe can trigger a local twitch response (LTR), which can reproduce symptoms of pain. This study will use a digital algometer to measure pressure pain threshold, which have been used by previous authors (Luan et al, 2019).

Most patients with MPS are treated by physiotherapists, physicians, chiropractors and osteopaths using trigger point injection, dry needling, acupuncture, ultrasound, stretches, deep frictional massages and taping (Galasso et al, 2020; Tough et al, 2009; Müller-Ehrenberg, 2005; Fernández-de-las-Peñas, et al, 2012). However, the most effective treatment for MPS is not known.

Radial shockwave is one of the most common and non-invasive treatments method with very few negative side effects, for musculoskeletal tissues such as MPS that normally are very difficult to treat (Watson, 2014). They are low to medium-energy pulses and their penetration depths are normally 0-6 cm ("0-2.3") (Watson, 2014). The therapeutic doses of radial shockwave ranges from low (up to 0.08mJ/mm2) to high (up to 0.63mJ/mm2) energy levels, and the number of treatment session repetitions is between 3 - 7 sessions (Watson, 2014). The number of shocks per session is usually between 1000 to 2500.

Some of the most strongly established therapeutic and biological effects of radial shockwave include mechanical stimulation, increased local blood flow that leads to tissue repair and regeneration by causing micro-functional and micro-structural changes, increase in cellular activity - release of substance P, prostaglandin E2 and tumour growth factor (TGF β), transient analgesic effect on afferent nerves and break down of calcific deposits (Watson, 2014; Wang, 2012). No evidence of serious tissue destruction at therapy level doses has been reported.

Some authors (Kiraly et al, 2018, Lee & Han, 2013; Gur et al, 2013, Cho et al, 2012) have demonstrated the efficacy of shockwave therapy to improve outcomes of pain and function in neck pain patients with MPS despite unclear pathophysiology. Despite these findings, recent systematic reviews (Yoo et al, 2020; Jun et al, 2021), found very low-level evidence to support its use for pain relief in patients with MPS in the neck in the short-term, due to the poor methodological qualities and small sample size. The authors therefore recommended the need for further large scale, good quality placebo-controlled trials in this area. Furthermore, previous studies (Manafnezhad et al, 2019; Gur et al, 2013; and Jeon et al, 2012) that have compared the effectiveness of shockwaves therapy have not done so with a true placebo. A truly appropriate placebo must be biologically inactive and psychologically credible-meaning it must be indistinguishable (by the patient) from real intervention (Vickers, 2002).

Further still, previous studies on the effect of shockwave therapy on MPS did not consider the experiences of patient regarding this intervention. Besides, to our knowledge and despite extensive literature search, no study has compared both the effectiveness of shockwave on MPS and the experiences of the patients receiving the treatment. This study will therefore investigate the effectiveness of radial shockwave therapy at reducing pain, disability and improving function in neck and upper back pain in patients MPS. It will also explore the experiences of patients receiving this treatment.

Aims of the Study Primary Aims

1. To determine the effectiveness of radial shockwave therapy compared to placebo for the treatment of patients with MPS in neck and upper back
2. To establish the experiences of patients with MPS in the neck and upper back receiving radial shockwave treatment

Research Question

1. Is radial shockwave therapy more effective at improving MPS in neck and upper back and compared to a placebo?
2. What are the experiences of patients with MPS in the neck and upper back receiving radial shockwave therapy?

METHODS

PHASE 1 METHODS Design: Quantitative - Randomised Controlled Trial This study will make use a two-arm, doubled-blind, randomised controlled design as defined by Hicks (1999), where the effects on dependent variables (neck and upper back pain and function) will be measured by manipulating two independent variables radial shockwave therapy and a placebo. RCTs are regarded as gold standard when evaluating the effectiveness of interventions because they enable us to be confident that a difference in outcome can be directly attributed to a difference in the treatments and not due to some other factors such as confounders (McGovern 2001). However, the experience of receiving such intervention of may play a role (Black 1996).

Study Setting This study will take place at the outpatient department of the Physical Rehabilitation, in King Faisal Specialist Hospital & Research Centre (KFSHRC). Prior to the study, presentations will be made to the Family Physicians in KFSHRC and the Physical Rehabilitation staff to inform them of the study. They will be provided with details regarding the rationale behind the study and the potential participants. Potential participants will be recruited from the outpatient of KFSHRC-Physical Rehabilitation Department.

Identification of Potential Participants Potential participants will be patients that have been referred to the Physical Rehabilitation service by the family physician and/or other specialists in KFSHRC with neck and/or upper back pain. At first appointment, a Physical Therapists (PT) will then identify them through a face-to-face assessment to determine if they have a diagnosis of MPS in the neck and or upper pain and would benefit from a radial shockwave therapy. A diagnosis of MPS will be made by the assessing PT according to the inclusion and exclusion criteria in table 1.

Clinicians Involvement in the Study The Principal Investigator and five out-patient PTs who are trained and experienced in the use of radial shockwave therapy will be involved in this study. The trained and experienced PT will be involved in consenting, assessing and treating the patients. The same PT would be involved in the patient's initial assessment and the baseline measurement. Subsequent appointments and rate of progression would be determined by this physiotherapist. Information about the eligibility criteria will be provided to all PTs to aid diagnosis and they will receive training on the study protocol.

Recruitment of Potential Participants When the first PT appointment is made to the patient, a separate envelope containing a letter of invitation to take part in the study will be given to them by the admin staff. The invitation pack will contain a Patient Information Sheet (PIS) and consent form (for the quantitative part and qualitative interview) (see Appendix 1). In the Patient Information Sheet (PIS), it is clearly stated that involvement in the study is voluntary, and that participants will be free to withdraw from the study at any time. Potential participants who are interested in taking part in the study but have further questions will be encouraged to contact the Principal Investigator via a study mobile number. The phone number will be provided in the PIS. Potential participants will be asked to read the PIS before attending their first PT appointment when they will have an opportunity to ask questions if they wish to participate, and will be asked to sign the consent forms. On arriving for their first PT appointment, potential participants who provide written informed consent and fulfil the eligibility criteria after being screened by the assessing PT will be recruited into the study. Participants who do not wish to participate, will receive standard PT treatment.

Randomisation Randomisation will be based on concealed random allocation using sealed opaque envelopes. Allocation concealment ensures that participants and clinicians cannot know or predict what the next patient and treatment allocation will be (Viera et al 2007). Assignment will be made by sequentially numbered, otherwise identical, sealed envelopes. Envelopes will be opaque and lined inside with carbon paper. Each envelope will contain a 2-inch by 2-inch paper with a written code A or B designating intervention (radial shockwave therapy) or control (placebo) respectively. Following the opening of each envelope, the admin staff will assign the patient to either the intervention or control group using the label A or B on the sealed envelope. Following notification of the randomisation result by the admin staff, the treating PT will assign the patient to treatment allocation using the label A or B on the sealed envelope. The patient will receive either the experimental treatment (radial shockwave therapy) if the envelope is labelled A, or they will receive the control treatment (placebo) if it is labelled B. This process will minimise systematic bias because it will ensure that there are no order or time effects; and the treating PTs have been trained in both methods.

During their first PT appointment, participants will be required to give informed consent. After consent is given and the participant meets selection criteria for the study, they will be randomised into radial shockwave group - A or control group - B (1:1 allocation ratio) using a computer generated randomization codes by the administration staff. Each envelope labelled A will be given a corresponding number code such as A1, A2, A3, etc will represent the radial shockwave therapy. Those labeled B will each have B1, B2, B3, etc will represent the placebo group. The patient's number code will represent whether they receive radial shockwave therapy or placebo by the treating PTs. This will correspond to the concealed random allocation design.

Outcome Measures and Follow up Baseline Assessment Baseline characteristics will include age, gender, duration of symptoms, current treatment analgesia and current treatment NSAIDS. It also includes the initial NPS, NDI, PPT and SF-12 scores See table 3 for details.

Follow-up Assessment Potential participants will be assessed three times during the study period, at 0 (baseline), 4, and 8 weeks. This will allow inferences to be drawn about immediate and short-term effects. The 8 weeks' timeframe is common in normal clinical practice. Follow-up assessments would be done by a Staff (who is not involved in the patient's treatment and blinded to the baseline measurement and group allocation), at 4 and 8 weeks. These timeframes are normal clinical practice and consistent with previous authors (Luan et al, 2019; Eftekharsadat et al, 2020).

Blinding The blinded assessor - a staff who can speak both English and Arabic Language (who is not involved in the patient's treatment and blinded to the baseline measurement and group allocation), will collect the outcomes at 4 and 8 weeks. Where necessary, response rate will also be facilitated through a call reminder of up to two occasions each time to ask if they wish to complete the questionnaires. The statistician conducting the primary data analysis will also be blinded to the group allocation.

Potential participants will be blinded to the treatment allocation. They will not know if they are receiving the experimental or placebo treatment. However, it is not possible for the treating PTs to be blinded to treatment allocation with this design because they already know what the experimental and placebo treatment is. However, they do not control which patient they treat because of the concealed random allocation of potential participants.

Loss to Follow-up This study is likely to last for 12 months' study, therefore, at 4 months a review of the rate of loss to follow-up will be undertaken to ensure that this does not affect the findings of the study. For example, if the rate of loss to follow-up is much higher in one group compared with the other, the researcher might consider over enrolling into that group. Patients who are lost to follow-up will be included in the analysis based on intention to treat (ITT).

Data and Treatment Fidelity Treating physiotherapists are skilled, trained and experienced in the management of MPS using radial shockwaves. To ensure procedural integrity of the study, the assessment and treatment given to potential participants from the RCT will be evaluated by the Principal Investigator (CO). Standardised training on the study procedure will also be provided to the treating physiotherapists to facilitate successfully delivery of both treatments (see Appendix 6). Administrative staff involved in the study will receive training on the study protocol. Some of the treatment sessions from both groups of the study will be observed, documented and feedback would be provided to the treating physiotherapists. The radial shockwave machines for this study would have passed their normal regular checks to ensure they are properly calibrated and working well. Participants will be randomly selected and interviews will be conducted 3 months after their initial treatment to get their views on the care they received.

Sample Size Calculations Sample size calculations will be based on works by Aktürk et al (2018) and Gur et al (2014). We estimated the minimal clinically important difference (MCID) to be a change in NPS of 2 points, at 90% power, with a statistical significance level of 5% and a standard deviation of 4.35 points. Using these figures, a sample of 100 participants is estimated for the study. However, to account for a 20% rate of loss at follow-up, this study will include 120 participants. Therefore, each study group will have 60 participants.

Non-Response and Intention to Treat Analysis Participants who withdraw from the study will be included in the analysis based on intention to treat (ITT). ITT analysis therefore helps to prevent two major issues such as noncompliance and missing data that are associated with RCT (Gupta 2011). The ITT analysis takes into account all randomised patients in the groups to which they were randomly assigned, regardless of their adherence with the entry criteria, treatment they actually received, and subsequent withdrawal from treatment or deviation from the study protocol (Kruse et al 2002; Fisher et al 1990).

Plan of Analysis All analyses will be undertaken on an intention to treat basis. All data will be analysed using the BM SPSS Statistics version 20 (SPSS Inc., Chicago, IL). Descriptive statistics such as mean age, gender and duration of symptoms will be used to describe patient's baseline characteristics. The results of the outcome measures will give a difference in scores from the baseline to 4 and 8 weeks. All analyses will be undertaken on an intention to treat basis. Normality will also be checked using the Sharipo-Wilk test since the sample size is 120. The chi-square test will be used to compare the distribution of categorical variables. We will use a paired sample t test for analysing within group difference, and independent sample t test for analyzing between group. A regression model will be used to evaluate the contribution of participant's baseline characteristics such as age, gender, symptom duration. Significance level is set at P ≤ 0.05 with a 95% confidence interval to detect a minimal clinically important difference of 2 points between the groups receiving shockwave therapy and placebo treatment.

Ethical Considerations Approval was obtained from the Research Ethics Committee (REC), King Faisal Specialist Hospital and Research Centre on 07 April 2022 (#2221047). Written informed consent, a prerequisite for study participation, would be obtained from all participants. Potential participants will be given the opportunity to determine if they want to participate in the study or not. The relevance of the research, including the possible risks and benefits, will be carefully explained to them. This is to enable participants to give informed consent based on an understanding that their participation in this research is voluntary.

Potential participants will be informed that they are not obliged to take part in the study and that failure to provide consent or withdrawal of consent without giving a reason will not affect the treatment that they will receive. All participants' details, as well as their comments, will be kept secure and confidential at all-times using a locked cabinet (with controlled access) and on a password protected computer. Any information they provide to Principal Investigator will be anonymised using pseudonyms and unique identifying numbers, so that it will not be possible to identify them. Dictaphone recordings of interviews will be destroyed once they have been transcribed and transcripts will be stored in a locked cabinet (with controlled access) and on a password protected computer.

No significant adverse reactions are anticipated in the study, but these will be monitored and recorded by department's ethics committee lead. Participants were informed that their Physician would be informed of their participation in the study and after obtaining consent from them to do so, the patient's Family Physician will be informed via a letter of their patient's participation in the study. If a participant is feeling distressed or uncomfortable during the trial, they will be advised to consult their Family Physician and will be excluded from the study, but any data collected up to that point will be included in the analysis.

Potential participants would be informed that there are not any direct personal benefits to them taking part in this study. However, the information derived from the study would help clinicians to know which of the two treatment methods is better in treating patients with MPS in the neck and upper back region in the future. Potential participants will be informed that they will be offered radial shockwave or placebo and each group will receive in addition the usual PT treatments associated with this condition. Both groups will receive the usual care including some exercise that is usually associated with MPS. However, all exercise will be performed at a speed and intensity that is within participant's own control.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19 and above
* Neck and or upper back pain localised the lateral or posterior neck and or upper back
* Palpable tenderness in the lateral or posterior neck and or upper back
* Trigger points in lateral or posterior neck and or upper back
* Able to give informed consent

Exclusion Criteria:

* Patients below 19 years of age
* History of:

  * Malignancy
  * Lung tissue
  * Haemophiliacs or patients on anticoagulant therapy
  * Visible tissue damage (skin petechiae & microvasculature disruption)
  * Metal implants - implanted cardiac stents & heart valves
  * Infection
  * Rheumatic, respiratory, cardiovascular diseases
  * Psychopathy
  * Disorders of the vestibular and visual systems
  * neck or shoulder surgery within a year,
  * Recent history steroid injections to myofascial trigger point
  * Pregnancy
* Diagnosed as:

  • Fibromyalgia, cervical radiculopathy or myelopathy
* Inability and unwillingness to continue study
* Failure to consent

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale (NPRS) | 12 weeks
  NPRS is a single 11-point numeric scale (with 0 as "no pain" and 10 as the "worse imaginable pain") to measure pain intensity in adults (Hawker 2011). It allows patients to measure their level of pain accordingly using a whole number (0-10 integers) that corresponds to their pain intensity (Rodriguez, 2001). The scale is considered reliable (accurate and consistent), responsive (ability to detect clinically significant changes) and valid (actually measures what it sets out to) (Hawker, 2011). Accordingly, a pain reduction of 2 points, or 30%, on the NPRS scores is defined as Minimal Clinically Important Difference (MCID) [Childs et al, 2005; Farrar et al, 2001]. The NPS is relatively easy to comprehend, and to apply, especially by patients with musculoskeletal disorders (Hawker, 2011).
Neck Disability Index (NDI) | 12 weeks
  It is the most commonly used self-rated disability score for assessing patients with neck pain Vernon & Mior (1991). It consists of ten domains: pain intensity, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation. Each question contains six answer choices, scored from 0 (no disability) to 5 (complete disability). All sections are then totalled. Scoring is reported on a 0-50 scale, 0 being the best possible score and 50 being the worst. The score can also be reported as a percentage (0-100%). The Minimum Detectable Change (90% confidence) is 5 points or 10% points Vernon & Mior (1991), and the MCID is in the range of 3.5-5.0 points (Pool et al, 2007).
Pressure pain threshold (PPT) | 12 weeks
  It will be measured using a digital algometer and pain score measurement will be performed with digital palpation. The algometer circular flat tip with 1.0 cm2 surface will be slowly pushed vertically to the skin over the trigger points until the participants interprets the compression on skin as pain sensation. The exerted pressure will be enlarged at a rate of 1 kg/cm2. Participants will be requested to inform the treating physiotherapist by saying "yes" when the pain is perceived. The measurements will be taken three times with 40 seconds intervals, and the mean average value will be taken (Fischer, 1998). A mean difference of 0.94 kg/cm2 in PPT was defined as MCID (Asiri et al, 2020).
SF12 - Quality of life (QoL) | 12 weeks
  Quality of life status will be evaluated using the short form (SF12), which is a shorter version of SF-36 questionnaire. The health survey (SF-12) questionnaire, consists of 12 items regarding the quality of life with respect to the physical and emotional aspects. Likert scales and yes/no options were used to assess function and wellbeing on this 12-item questionnaire. To score the SF-12, scales are standardized with a scoring algorithm to obtain a score ranging from 0 to 100. Higher scores indicate better health status. It is one of the most widely used patient report outcome with well documented high validity, reliability, and responsiveness rate among many groups varying by age, sex, socio-economic status, geographical region, and clinical conditions (Ware et al, 2000).

CONTACTS AND LOCATIONS:
Locations (1):
- Physical Rehabilitation Department, King Faisal Specialist Hospital & Research Centre, Riyadh, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alvarez DJ, Rockwell PG. Trigger points: diagnosis and management. Am Fam Physician. 2002 Feb 15;65(4):653-60. PMID 11871683
- [Background] Akturk S, Kaya A, Cetintas D, Akgol G, Gulkesen A, Kal GA, Gucer T. Comparision of the effectiveness of ESWT and ultrasound treatments in myofascial pain syndrome: randomized, sham-controlled study. J Phys Ther Sci. 2018 Mar;30(3):448-453. doi: 10.1589/jpts.30.448. Epub 2018 Mar 2. PMID 29581669
- [Background] Asiri F, Tedla JS, D Alshahrani MS, Ahmed I, Reddy RS, Gular K. Effects of patient-specific three-dimensional lumbar traction on pain and functional disability in patients with lumbar intervertebral disc prolapse. Niger J Clin Pract. 2020 Apr;23(4):498-502. doi: 10.4103/njcp.njcp_285_19. PMID 32246656
- [Background] Black N. Why we need observational studies to evaluate the effectiveness of health care. BMJ. 1996 May 11;312(7040):1215-8. doi: 10.1136/bmj.312.7040.1215. PMID 8634569
- [Background] Cho YS, Park SJ, Jang SH, Choi YC, Lee JH, Kim JS. (2012). Effects of the combined treatment of extracorporeal shock wave therapy (ESWT) and stabilization exercises on pain and functions of patients with myofascial pain syndrome. J Phys Ther Sci; 24:1319-23.
- [Background] Childs JD, Piva SR, Fritz JM. Responsiveness of the numeric pain rating scale in patients with low back pain. Spine (Phila Pa 1976). 2005 Jun 1;30(11):1331-4. doi: 10.1097/01.brs.0000164099.92112.29. PMID 15928561
- [Background] Coombes BK, Bisset L, Vicenzino B. A new integrative model of lateral epicondylalgia. Br J Sports Med. 2009 Apr;43(4):252-8. doi: 10.1136/bjsm.2008.052738. Epub 2008 Dec 2. PMID 19050004
- [Background] Eftekharsadat B, Fasaie N, Golalizadeh D, Babaei-Ghazani A, Jahanjou F, Eslampoor Y, Dolatkhah N. Comparison of efficacy of corticosteroid injection versus extracorporeal shock wave therapy on inferior trigger points in the quadratus lumborum muscle: a randomized clinical trial. BMC Musculoskelet Disord. 2020 Oct 19;21(1):695. doi: 10.1186/s12891-020-03714-3. PMID 33076888
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728
- [Background] Fernandez-de-las-Penas C, Grobli C, Ortega-Santiago R, Fischer CS, Boesch D, Froidevaux P, Stocker L, Weissmann R, Gonzalez-Iglesias J. Referred pain from myofascial trigger points in head, neck, shoulder, and arm muscles reproduces pain symptoms in blue-collar (manual) and white-collar (office) workers. Clin J Pain. 2012 Jul;28(6):511-8. doi: 10.1097/AJP.0b013e31823984e2. PMID 22673484
- [Background] Fischer AA. Documentation of myofascial trigger points. Arch Phys Med Rehabil. 1988 Apr;69(4):286-91. PMID 3281631
- [Background] Fisher LD, Dixon DO, Herson J, Frankowski RK, Hearron MS & Peace KE (1990) Intention to treat in clinical trials. In: Peace KE, editor. Statistical issues in drug research and development. New York: Marcel Dekker.
- [Background] Fleckenstein J, Zaps D, Ruger LJ, Lehmeyer L, Freiberg F, Lang PM, Irnich D. Discrepancy between prevalence and perceived effectiveness of treatment methods in myofascial pain syndrome: results of a cross-sectional, nationwide survey. BMC Musculoskelet Disord. 2010 Feb 11;11:32. doi: 10.1186/1471-2474-11-32. PMID 20149248
- [Background] Galasso A, Urits I, An D, Nguyen D, Borchart M, Yazdi C, Manchikanti L, Kaye RJ, Kaye AD, Mancuso KF, Viswanath O. A Comprehensive Review of the Treatment and Management of Myofascial Pain Syndrome. Curr Pain Headache Rep. 2020 Jun 27;24(8):43. doi: 10.1007/s11916-020-00877-5. PMID 32594264
- [Background] Gaskin DJ, Richard P. The economic costs of pain in the United States. J Pain. 2012 Aug;13(8):715-24. doi: 10.1016/j.jpain.2012.03.009. Epub 2012 May 16. PMID 22607834
- [Background] Gupta SK. Intention-to-treat concept: A review. Perspect Clin Res. 2011 Jul;2(3):109-12. doi: 10.4103/2229-3485.83221. PMID 21897887
- [Background] Gur, A., Koca, I., Karagullu, H., Altindag, O., & Madenci, E. (2013). Comparison of the efficacy of ultrasound and extracorporeal shock wave therapies in patients with myofascial pain syndrome: a randomized controlled study. Journal of musculoskeletal Pain, 21(3), 210-216. DOI: 10.3109/10582452.2013.828824.
- [Background] Green S, Buchbinder R, Hetrick S. Physiotherapy interventions for shoulder pain. Cochrane Database Syst Rev. 2003;2003(2):CD004258. doi: 10.1002/14651858.CD004258. PMID 12804509
- [Background] Haddad C, Sacre H, Obeid S, Salameh P, Hallit S. Validation of the Arabic version of the "12-item short-form health survey" (SF-12) in a sample of Lebanese adults. Arch Public Health. 2021 Apr 23;79(1):56. doi: 10.1186/s13690-021-00579-3. PMID 33892801
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Jeon JH, Jung YJ, Lee JY, Choi JS, Mun JH, Park WY, Seo CH, Jang KU. The effect of extracorporeal shock wave therapy on myofascial pain syndrome. Ann Rehabil Med. 2012 Oct;36(5):665-74. doi: 10.5535/arm.2012.36.5.665. Epub 2012 Oct 31. PMID 23185731
- [Background] Jun JH, Park GY, Chae CS, Suh DC. The Effect of Extracorporeal Shock Wave Therapy on Pain Intensity and Neck Disability for Patients With Myofascial Pain Syndrome in the Neck and Shoulder: A Meta-Analysis of Randomized Controlled Trials. Am J Phys Med Rehabil. 2021 Feb 1;100(2):120-129. doi: 10.1097/PHM.0000000000001493. PMID 32520797
- [Background] Kiraly M, Bender T, Hodosi K. Comparative study of shockwave therapy and low-level laser therapy effects in patients with myofascial pain syndrome of the trapezius. Rheumatol Int. 2018 Nov;38(11):2045-2052. doi: 10.1007/s00296-018-4134-x. Epub 2018 Aug 31. PMID 30171341
- [Background] Kruse RL, Alper BS, Reust C, Stevermer JJ, Shannon S, Williams RH. Intention-to-treat analysis: who is in? Who is out? J Fam Pract. 2002 Nov;51(11):969-71. PMID 12485553
- [Background] Lauche R, Langhorst J, Dobos GJ, Cramer H. Clinically meaningful differences in pain, disability and quality of life for chronic nonspecific neck pain - a reanalysis of 4 randomized controlled trials of cupping therapy. Complement Ther Med. 2013 Aug;21(4):342-7. doi: 10.1016/j.ctim.2013.04.005. Epub 2013 May 25. PMID 23876565
- [Background] Lee, J. H., & Han, E. Y. (2013). A comparison of the effects of PNF, ESWT, and TPI on pain and function of patients with myofascial pain syndrome. Journal of Physical Therapy Science, 25(3), 341-344.
- [Background] Li X, Wang R, Xing X, Shi X, Tian J, Zhang J, Ge L, Zhang J, Li L, Yang K. Acupuncture for Myofascial Pain Syndrome: A Network Meta-Analysis of 33 Randomized Controlled Trials. Pain Physician. 2017 Sep;20(6):E883-E902. PMID 28934793
- [Background] Luan S, Zhu ZM, Ruan JL, Lin CN, Ke SJ, Xin WJ, Liu CC, Wu SL, Ma C. Randomized Trial on Comparison of the Efficacy of Extracorporeal Shock Wave Therapy and Dry Needling in Myofascial Trigger Points. Am J Phys Med Rehabil. 2019 Aug;98(8):677-684. doi: 10.1097/PHM.0000000000001173. PMID 31318748
- [Background] Manafnezhad J, Salahzadeh Z, Salimi M, Ghaderi F, Ghojazadeh M. The effects of shock wave and dry needling on active trigger points of upper trapezius muscle in patients with non-specific neck pain: A randomized clinical trial. J Back Musculoskelet Rehabil. 2019;32(5):811-818. doi: 10.3233/BMR-181289. PMID 30883334
- [Background] McGovern, D. P. B. (2001). Randomized controlled trials. In: McGovern DPB, Valori RM, Summerskill WSM, eds. Key topics in evidence based medicine. Oxford: BIOS Scientific Publishers: 26 - 9.
- [Background] Müller-Ehrenberg, H., & Licht, G. (2005). Diagnosis and therapy of myofascial pain syndrome with focused shock waves (ESWT). Med Orthop Tech, 5, 1-6.
- [Background] Pool JJ, Ostelo RW, Hoving JL, Bouter LM, de Vet HC. Minimal clinically important change of the Neck Disability Index and the Numerical Rating Scale for patients with neck pain. Spine (Phila Pa 1976). 2007 Dec 15;32(26):3047-51. doi: 10.1097/BRS.0b013e31815cf75b. PMID 18091500
- [Background] Rodriguez CS. Pain measurement in the elderly: a review. Pain Manag Nurs. 2001 Jun;2(2):38-46. doi: 10.1053/jpmn.2001.23746. PMID 11706769
- [Background] Sciotti VM, Mittak VL, DiMarco L, Ford LM, Plezbert J, Santipadri E, Wigglesworth J, Ball K. Clinical precision of myofascial trigger point location in the trapezius muscle. Pain. 2001 Sep;93(3):259-266. doi: 10.1016/S0304-3959(01)00325-6. PMID 11514085
- [Background] Simons, D G. (1996) Clinical and Etiological Update of Myofascial Pain from Trigger Points, Journal of Musculoskeletal Pain, 4:1-2, 93-122, DOI: 10.1300/J094v04n01_07.
- [Background] Travell, J. G., & Simons, D. G. (1999). Myofascial Pain and Dysfunction: The Trigger Point Manual. 2nd ed. (Vol 1). Baltimore, MD: Williams and Wilkins.
- [Background] Tough EA, White AR, Cummings TM, Richards SH, Campbell JL. Acupuncture and dry needling in the management of myofascial trigger point pain: a systematic review and meta-analysis of randomised controlled trials. Eur J Pain. 2009 Jan;13(1):3-10. doi: 10.1016/j.ejpain.2008.02.006. Epub 2008 Apr 18. PMID 18395479
- [Background] Vernon H, Mior S. The Neck Disability Index: a study of reliability and validity. J Manipulative Physiol Ther. 1991 Sep;14(7):409-15. PMID 1834753
- [Background] Vickers AJ. Placebo controls in randomized trials of acupuncture. Eval Health Prof. 2002 Dec;25(4):421-35. doi: 10.1177/0163278702238055. PMID 12449085
- [Background] Viera AJ, Bangdiwala SI. Eliminating bias in randomized controlled trials: importance of allocation concealment and masking. Fam Med. 2007 Feb;39(2):132-7. PMID 17273956
- [Background] Ware JE Jr. SF-36 health survey update. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3130-9. doi: 10.1097/00007632-200012150-00008. No abstract available. PMID 11124729
- [Background] Watson, P (2014) Shockwave therapy, available online at: shockwave Prof Time Watson.pdf.
- [Background] Wang CJ. Extracorporeal shockwave therapy in musculoskeletal disorders. J Orthop Surg Res. 2012 Mar 20;7:11. doi: 10.1186/1749-799X-7-11. PMID 22433113
- [Background] Yoo JI, Oh MK, Chun SW, Lee SU, Lee CH. The effect of focused extracorporeal shock wave therapy on myofascial pain syndrome of trapezius: A systematic review and meta-analysis. Medicine (Baltimore). 2020 Feb;99(7):e19085. doi: 10.1097/MD.0000000000019085. PMID 32049811
- [Derived] Ogbeivor C, AlMubarak H, Akomolafe T, Alkahtani H, AlMugizel H, Marin I, Aldosari H, Aldhwayan N, Mohamed G, Alobthani K. The effectiveness of radial shockwave therapy on myofascial pain syndrome: a two-armed, randomized double-blind placebo-controlled trial. BMC Musculoskelet Disord. 2025 Apr 24;26(1):413. doi: 10.1186/s12891-025-08659-z. PMID 40275291